CLINICAL TRIAL: NCT05979129
Title: Comparing the Incidence of Gastric Insufflation During Facemask Ventilation at Different Levels of End-expiratory Pressure During Induction of Anesthesia in Obese Patients: a Randomized Controlled Study
Brief Title: Gastric Insufflation During Facemask Ventilation at Different Levels of End-expiratory Pressure in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Maha Mostafa Ahmad, MD, assistant professor, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MD-65-2022
Record Dates: First submitted 2023-07-30; First posted 2023-08-07 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Gastric Insufflation; Face-mask Ventilation; Obese; Positive End Expiratory Pressure
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ZEEP group (Active Comparator)
  Interventions: Other: zero PEEP
- Low PEEP (Active Comparator)
  Interventions: Other: low PEEP
- High PEEP (Active Comparator)
  Interventions: Other: high PEEP

INTERVENTIONS:
Other: zero PEEP — zero end-expiratory pressure during face mask ventilation
  Arms: ZEEP group
Other: low PEEP — 4 cmH2O PEEP during mask ventilation
  Arms: Low PEEP
Other: high PEEP — 8 cmH2O PEEP during mask ventilation
  Arms: High PEEP

SUMMARY:
Gastric insufflation occurs when the inspiratory pressure exceeds the lower esophageal sphincter pressure. Thus, it is desirable to avoid excessive positive pressure during mask ventilation after induction of anesthesia and keeping the inspiratory pressure <15-20 cmH2O.In patients with obesity the lower compliance of the respiratory system usually requires higher inspiratory pressures to maintain adequate ventilation making these patients more prone to gastric insufflation. This high risk of gastric insufflation can be aggravated by the use of positive end-expiratory pressure (PEEP) which is recommended to avoid lung atelectasis. The application of PEEP during mask ventilation increases the risk of gastric insufflation as it reduces the pressure threshold at which gastric insufflation occur The optimum ventilatory strategy during mask ventilation should achieve the balance between adequate lung ventilation and avoiding gastric insufflation. In obese patients, it is not clear whether the use of PEEP during mask ventilation would increase the risk of gastric insufflation or not.

We hypothesize that using zero end-expiratory pressure (ZEEP) or low PEEP during mask ventilation would reduce the risk of gastric insufflation in comparison to high PEEP.

DETAILED DESCRIPTION:
Upon arrival to the operating room, routine monitors (electrocardiogram, pulse oximetry, and non-invasive blood pressure monitor) will be applied, intravenous line will be secured. End-tidal CO2 monitoring will be initiated after induction of general anesthesia and starting face-mask ventilation. All patients will be positioned in the ramped position (achieved by elevation of the head and shoulders till achieving alignment of sternal notch and external auditory meatus). Preoxygenation will be achieved by pressure support ventilation with 5 cmH2O and FiO2 of 0.8 without PEEP for three minutes. Induction of anesthesia will be achieved using fentanyl (2 mcg/Kg lean body weight), propofol (2 mg/Kg lean body weight), and rocuronium (0.6 mg/Kg ideal body weight). After loss of verbal response, mask ventilation will be achieved by appropriate size face mask and oropharyngeal airway with 100% oxygen and double hand jaw thrust head tilt maneuver. The included patients will be receiving volume-controlled ventilation adjusted to deliver tidal volume of 8-10 mL/kg (ideal body weight), at I:E ratio of 1:2, inspiratory pause of 0.5 s, respiratory rate of 12 breath per minute, FiO2 of 0.8.

The 3 study groups will receive the planned ventilatory strategy for 120 seconds.

Assessment gastric insufflation during mask ventilation will be achieved by ultrasound assessment of gastric antrum (at the sagittal plane between left lobe of the liver and pancreas at level of the aorta). Gastric antral cross-sectional area (CSA) [ (longitudinal diameter) X (anteroposterior diameter) X π /4] will be assessed in between contractions before face mask ventilation and after insertion of endotracheal tube. [9] The proportion of change in the CSA will be calculated as (delta CSA %= [CSA after intubation - baseline CSA] / baseline CSA X 100). Significant gastric insufflation will be identified if the CSA increased by > 30% after endotracheal intubation in relation to the baseline.

Intermittent gastric auscultation will be performed during mask ventilation at 30, 60, 90, 120 seconds by a blinded investigator (the presence of gastric insufflation will be defined as a gurgling sound).

ELIGIBILITY:
Inclusion Criteria:

* adult patients,
* with American Society of Anesthesiologists physical status II,
* body mass index >35 kg/m2,
* scheduled for elective surgery under general anesthesia.

Exclusion Criteria:

* Patients at increased risk of difficult mask ventilation: Mallampati classification >2, presence of beard, limited neck extension, limited jaw protrusion, patients with history of obstructive sleep apnea or STOP-Bang score>2
* Patients at risk of aspiration or history of esophageal reflux.
* Patients with craniofacial anomalies, and pregnant patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2023-08-06 (Actual); Primary Completion 2024-04-28 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Change in gastric cross sectional area more than 30% | 1 minute before preoxygenation and 1 minute after intubation
  number of patients with increase in percentage of change in gastric cross sectional area by more than 30%

SECONDARY OUTCOMES:
gastric cross sectional area | 1 minute before preoxygenation and 1 minute after intubation
  gastric cross sectional area measured by ultrasonography in cm2
percentage of change in gastric cross sectional area | 1 minute before preoxygenation and 1 minute after intubation
  gastric cross sectional area after intubation divided by gastric cross sectional area before preoxygenation %
tidal volume | 30 seconds until 120 seconds after induction of anesthesia
  mL/kg
end-tidal CO2 | 30 seconds until 120 seconds after induction of anesthesia
  mmHg
Peak airway pressure | 30 seconds until 120 seconds after induction of anesthesia
  mmHg
Gastric insufflation | 30 seconds until 120 seconds after induction of anesthesia
  incidence of gastric insufflation by auscultation

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alaini Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data from this study will be available from PI upon reasonable request

REFERENCES:
- [Derived] Mostafa M, Hasanin A, Zakaria MM, Kandel H, Hamimy W, Abougabal A, Elshal MM. Comparing the effect of three levels of end-expiratory pressure during facemask ventilation on gastric insufflation in patients with obesity: a randomized controlled trial. J Anesth. 2025 Dec;39(6):887-895. doi: 10.1007/s00540-025-03531-9. Epub 2025 Jun 30. PMID 40586940